CLINICAL TRIAL: NCT01784484
Title: Screening for Liver Fibrosis by Using Non-invasive Methods ( Fibro Scan) in Patients With Elevated Liver Enzymes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assy Nimer (Other Government)
Responsible Party: Sponsor-Investigator, Assy Nimer, Prof. Assy Nimer, Ziv Hospital
Organization: Ziv Hospital (Other Government)
Other Study IDs: 0058-12-ZIV
Record Dates: First submitted 2013-01-23; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Elevated Liver Enzymes

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with abnormal liver enzymnes
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
BACKGROUND: Fibrosis assessment by Transient Elastography or Fibro scan is validated in chronic hepatitis C, however limited data are available in chronic hepatitis B and in non alcoholic fatty liver disease (NAFLD). AIMS: Document the prevalence and severity of fibrosis in patients with different chronic liver disease (elevated liver enzymes) who are being followed up in the liver unit and to find associated factors with significant fibrosis and cirrhosis at ziv medical center, Safed,Bar Ilan University. Israel. METHODS: Fibro scan will be performed to all patients with abnormal liver enzymnes who attend the liver clinic. Liver stiffness measurement, age, gender, BMI, will be measured. Questionaire on soft drink consumption, Coffee drinking, use of herbs, and a history of cancer or heart disease will be distributed. Expected RESULTS: we expect that the liver stiffness (normal 1-6 Kpa) will be higher in NAFLD patients than in viral hepatitis patients for the same age ,same BMI, and the same duration of disease. More over, we expect serum aspartate aminotransferase (AST) values will emerge as the most important independent predictive variable of fibrosis and not serum ALT. A significant correlations between soft drink and coffee consumption with the extent of liver fibrosis is also expected. CONCLUSIONS: This prospective study will confirm that screening patients with elevated liver enzymes is beneficial and detect earlier the presence of liver fibrosis mainly in patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* More than 18 years of age
* Patients with elevated liver enzymes
* Written informed consent

Exclusion Criteria:

* Patients refusing to participate to the study and to provide written informed consent
* clotting disorder
* ongoing treatment with anti-coagulant or anti-aggregant
* advanced or decompensated cirrhosis (Child-Pugh class C)
* hepatocellular carcinoma
* other cancer
* history of surgery for brain aneurysm
* pace maker or defibrillator
* ocular metal foreign body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abnormal liver enzymnes who attend the liver clinic
Sampling Method: Non-Probability Sample
Dates: Start 2013-02; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
liver stiffness | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel, Israel